CLINICAL TRIAL: NCT06390033
Title: Biomechanical Study of Different Prostheses for Unilateral Transtibial Amputees During Indoor and Outdoor Activities
Status: Completed | Type: Observational
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, YICK Kit Lun, Professor, The Hong Kong Polytechnic University
Other Study IDs: ITS/133/21
Record Dates: First submitted 2024-03-13; First posted 2024-04-29 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2024-04

CONDITIONS: Amputation; Prosthesis User
Keywords: unilateral transtibial amputee; low-cost prosthetic foot; elevated activities; biomechanical study

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- K2 or above prosthesis: Unilateral transtibial amputees will engage in both indoor and outdoor activities, utilizing their own prosthesis (control).
  Interventions: Device: Prosthetic foot
- A low-cost prosthesis: Unilateral transtibial amputees will engage in both indoor and outdoor activities, utilizing an experimental prosthesis
  Interventions: Device: Prosthetic foot

INTERVENTIONS:
Device: Prosthetic foot — Experimental prosthetic foot.

SUMMARY:
The goal of this observational study is to evaluate and compare the performance of two prosthetic feet for unilateral transtibial amputees during both indoor and outdoor activities. The main research questions aim to answer are:

1. Can a low-cost prosthetic foot enhance gait mechanics and physical performance in individuals who have undergone traumatic unilateral transtibial amputation, as compared to the traditional K2 - K3 prosthetic feet currently available on the market, during both indoor and outdoor activities?
2. Can the low-cost prosthetic foot meet user satisfaction levels after traumatic unilateral transtibial amputation, when compared to the traditional K2 - K3 prosthetic foot on the market?

Participants will be asked to do

1. Prior to the commencement of the experiment, a professional prosthetist and orthotist will conduct all fitting and alignment procedures for the transtibial amputees. Participants will then be given a two to three-week period to train and acclimate to the individual socket alignment and prosthetic foot.
2. Participants are asked to refrain from consuming caffeine or any stimulants for 24 hours before the tests.
3. Participants will be required to perform the Berg Balance Test.
4. Participants will undergo a series of clinical tests, including: 1) Time to Go Up (measured in seconds), 2) Four Square Step Test (measured in seconds), 3) 10-Meter Walk Test (measured in seconds), 4) Eye Close Standing, 5) Tandem Test, and 6) Functional Reach Test. Each test will be conducted three times. The test items of 4) and 5) will be performed on a force plate (Bertect, Ohio, USA) with dimensions of 400 x 600 mm and a capturing frequency of 1,000 Hz.
5. Participants will be asked to walk on a force plate (AMTI, Advanced Mechanical Technology, Inc., Watertown, USA) at a fixed walking speed of 1.11 ± 0.11m/s, allowing the foot to land naturally on the force plate. Five trials of the gait cycle with a clean foot will be used for analysis.
6. Participants will perform the Counter Movement Jump Test three times with maximum effort on the force plate (Bertect, Ohio, USA), which will be performed without a hand swing.
7. Participants will be asked to perform a 2-minute walking test on flat concrete ground, stairs, and a ramp, respectively.
8. Finally, participants will be asked to complete the Locomotion Capabilities Index questionnaire.

DETAILED DESCRIPTION:
Thirty-nine passive-reflective markers of 14 mm in diameter were placed on the participant (Figure 1) according to the landmarks set of the plug-in full body model. An 8-camera motion capturing system (VICON, Nexus 2.0 Inc., Oxford, UK) and 2 force plates (AMTI, Advanced Mechanical Technology, Inc., Watertown, USA) mounted under the walkway were utilized for gait analysis and recorded 100 frames per second simultaneously. All the systems were calibrated before the experiment.

ELIGIBILITY:
Inclusion Criteria:

* unilateral transtibial amputees,
* with more than 12 months of experience using a prosthesis,
* with a K2 prosthesis or above,
* be able to walk continuously unaided with the prosthetic foot for at least 20 minutes.

Exclusion Criteria:

* with a short or an injured residual limb,
* pregnant,
* any neurological or musculoskeletal diseases,
* have a record of active endocarditis and acute myocarditis/pericarditis,
* experience ongoing unstable angina,
* have uncontrolled cardiac arrhythmia with hemodynamic compromise,
* have had a recent stroke or transient ischemic attack,
* have high blood pressure, etc.

Ages: 36 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Six unilateral transtibial amputees (two females and four males) (age: (mean ± SD) 52.5 ± 12.1 years; height: 170.5 ± 10.5 cm; weight: 71.5 ± 6.5 kg; years using a prosthetic: 31 ± 10.8 years) were recruited in this study.
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Basic mobility function with two prostheses by Berg Balance Test | up to 12 weeks
  Participants will be invited to visit the laboratory twice to participate in two prostheses will be compared by conducting Berg Balance Test including 14 items, each item is graded using a 5-point ordinal scale ranging from 0 to 4. 0-20 indicates high fall risk, 21-40 indicates medium fall risk, 41-56 indicates low fall risk.
Basic mobility function with two prostheses by Time to Go Up | up to 12 weeks
  Participants will be invited to visit the laboratory twice to participate in two prostheses will be compared by conducting Time to Go Up (seconds), including stand up from chair, walk 3 meters, turn around and back, then sit. Longer than 13.5 seconds indicates high risk of fall.
Basic mobility function with two prostheses by Four Square Step Test | up to 12 weeks
  Participants will be invited to visit the laboratory twice to participate in two prostheses will be compared by conducting Four Square Step Test (seconds).
Basic mobility function with two prostheses by 10-meter Walk Test | up to 12 weeks
  Participants will be invited to visit the laboratory twice to participate in two prostheses will be compared by conducting 10-Meter Walk Test (m/s).
Stability index with two prostheses by Eye Close Standing | up to 12 weeks
  Participants will be invited to the laboratory twice to participate in an experiment. In each session, they will be required to perform the Eye Close Standing on a force plate (Bertect, Ohio, USA). The test will be conducted three times, with each attempt lasting 30 seconds. Participants will perform the task using either a low-cost prosthesis or their own prosthetic foot. The averaged anterior-posterior stability index (mm), and medial-lateral stability index (mm) will be calculated automatically by Noraxon software for each task to assess the ability of maintaining posture stability with two prostheses.
Stability index with two prostheses by Tandem Test | up to 12 weeks
  Participants will be invited to the laboratory twice to participate in an experiment. In each session, they will be required to perform the Tandem Test on a force plate (Bertect, Ohio, USA). The test will be conducted three times, with each attempt lasting 30 seconds. Participants will perform the task using either a low-cost prosthesis or their own prosthetic foot. The averaged anterior-posterior stability index (mm), and medial-lateral stability index (mm) will be calculated automatically by Noraxon software for each task to assess the ability of maintaining posture stability with two prostheses.
Functional Reach Test | up to 12 weeks
  Participants will move from the vertical standing position to the maximum lean forward position, with the feet firmly placed on the floor with either prosthetic foot for three times. The averaged distance (cm) with two prostheses will be compared.
Gait analysis with two prostheses | up to 12 weeks
  For collecting the kinematic and kinetic data for gait analysis, thirty-nine passive-reflective markers were placed on the participant according to the landmarks set of the plug-in full body model. An 8-camera motion capturing system (VICON, Nexus 2.0 Inc., Oxford, UK) and 2 force plates (AMTI, Advanced Mechanical Technology, Inc., Watertown, USA) mounted under the walkway were recorded 100 frames per second simultaneously. All the systems were calibrated before the experiment. Participants will be asked to walk on a force plate (AMTI, Advanced Mechanical Technology, Inc., Watertown, USA) at a fixed walking speed of 1.11 ± 0.11m/s, allowing the foot to land naturally on the force plate. Five trials of the gait cycle with a clean foot will be used for analysis.
Jump feasibility with two prostheses | up to 12 weeks
  Participants will be invited to visit the laboratory twice to participate in an experiment. During each visit, they will be asked to perform the countermovement jump on the force plate (Bertect, Ohio, USA) for three times, using either a low-cost prosthesis or their own prosthetic foot. The average of three times jump height, vertical ground reaction force during different jump phases with two different prostheses will be compared.
Subjective evaluation by Locomotion Capabilities Index questionnaire | up to 12 weeks
  Participants will be asked to complete the Locomotion Capabilities Index questionnaire including 14 items, each item is rated with a 5-level scale. 0 indicates unable to perform, 4 indicates no difficulty.

CONTACTS AND LOCATIONS:
Overall Officials: Kit-lun Yick, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Kowloon, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
IPD data related to this project will be only for publication purposes.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 30 June 2023 to 30 April, 2024
Access Criteria: IPD data related to this project will be only shared through publication.

REFERENCES:
- [Background] Kent JA, Stergiou N, Wurdeman SR. Dynamic balance changes within three weeks of fitting a new prosthetic foot component. Gait Posture. 2017 Oct;58:23-29. doi: 10.1016/j.gaitpost.2017.07.003. Epub 2017 Jul 5. PMID 28704685
- [Background] Pickenbrock HM, Diel A, Zapf A. A comparison between the Static Balance Test and the Berg Balance Scale: validity, reliability, and comparative resource use. Clin Rehabil. 2016 Mar;30(3):288-93. doi: 10.1177/0269215515578297. Epub 2015 Mar 23. PMID 25802425
- [Background] Franchignoni F, Orlandini D, Ferriero G, Moscato TA. Reliability, validity, and responsiveness of the locomotor capabilities index in adults with lower-limb amputation undergoing prosthetic training. Arch Phys Med Rehabil. 2004 May;85(5):743-8. doi: 10.1016/j.apmr.2003.06.010. PMID 15129398
- [Background] Segal AD, Orendurff MS, Klute GK, McDowell ML, Pecoraro JA, Shofer J, Czerniecki JM. Kinematic and kinetic comparisons of transfemoral amputee gait using C-Leg and Mauch SNS prosthetic knees. J Rehabil Res Dev. 2006 Nov-Dec;43(7):857-70. doi: 10.1682/jrrd.2005.09.0147. PMID 17436172
- [Background] Shi QQ, Yick KL, Wu J, Huang X, Tse CY, Chan MK. A Scientometric Analysis and Visualization of Prosthetic Foot Research Work: 2000 to 2022. Bioengineering (Basel). 2023 Sep 28;10(10):1138. doi: 10.3390/bioengineering10101138. PMID 37892868
- [Background] Arifin N, Abu Osman NA, Ali S, Wan Abas WA. The effects of prosthetic foot type and visual alteration on postural steadiness in below-knee amputees. Biomed Eng Online. 2014 Mar 5;13(1):23. doi: 10.1186/1475-925X-13-23. PMID 24597518
- [Background] Batten HR, McPhail SM, Mandrusiak AM, Varghese PN, Kuys SS. Gait speed as an indicator of prosthetic walking potential following lower limb amputation. Prosthet Orthot Int. 2019 Apr;43(2):196-203. doi: 10.1177/0309364618792723. Epub 2018 Aug 16. PMID 30112982
- [Background] Berg KO, Wood-Dauphinee SL, Williams JI, Maki B. Measuring balance in the elderly: validation of an instrument. Can J Public Health. 1992 Jul-Aug;83 Suppl 2:S7-11. PMID 1468055
- [Background] Dite W, Temple VA. A clinical test of stepping and change of direction to identify multiple falling older adults. Arch Phys Med Rehabil. 2002 Nov;83(11):1566-71. doi: 10.1053/apmr.2002.35469. PMID 12422327
- [Background] Gremeaux V, Damak S, Troisgros O, Feki A, Laroche D, Perennou D, Benaim C, Casillas JM. Selecting a test for the clinical assessment of balance and walking capacity at the definitive fitting state after unilateral amputation: a comparative study. Prosthet Orthot Int. 2012 Dec;36(4):415-22. doi: 10.1177/0309364612437904. Epub 2012 Mar 2. PMID 22389424
- [Background] Shumway-Cook A, Brauer S, Woollacott M. Predicting the probability for falls in community-dwelling older adults using the Timed Up & Go Test. Phys Ther. 2000 Sep;80(9):896-903. PMID 10960937